CLINICAL TRIAL: NCT04676763
Title: An Open Label, Single Centre, Enabling Study to Investigate the Optimum Method for Use of Intradermal Substance P as a Challenge Agent in Healthy Participants
Brief Title: Substance P Challenge in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 213224
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Skin Diseases
Keywords: Substance P; Wheal response; Flare response; Skin challenge
MeSH Terms: conditions — Skin Diseases | interventions — Substance P; Saline Solution; Histamine

STUDY DESIGN:
Intervention Model Description: Parts 1 and 2 will run sequentially. Part 1 will include 1 challenge visit; Part 2 will include two challenge visits.
Masking Description: It is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Substance P challenge in Part 1 (Experimental): Eligible participants will receive control challenge with saline and histamine, followed by challenge with ascending concentrations of Substance P. Part 1 will include a single challenge visit.
  Interventions: Drug: Substance P; Drug: Normal Saline; Drug: Histamine
- Substance P challenge in Part 2 (Experimental): Eligible participants will receive control challenge with saline and histamine, followed by challenge with ascending concentrations of Substance P. Part 2 will include two challenge visits.
  Interventions: Drug: Substance P; Drug: Normal Saline; Drug: Histamine

INTERVENTIONS:
Drug: Substance P — Participants will receive Substance P
Drug: Normal Saline — Participants will receive normal saline as Negative control
Drug: Histamine — Participants will receive histamine as Positive control

SUMMARY:
The objectives of this enabling study are to characterize the wheal and flare responses over time following skin challenges with ascending concentrations of Substance P. This will be a 2-part study: Part 1 will aid in the understanding of the wheal and flare responses following Substance P. Part 2 will investigate the variability of the responses. Participants may be enrolled into Part 1 or Part 2, not both.

ELIGIBILITY:
Inclusion criteria:

* 18 to 50 years of age inclusive.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, ECGs and vital signs.
* Participants who responded positive to histamine skin prick test and negative to saline injection at screening.
* Participants with Fitzpatrick skin type I-II (Caucasian).
* Body weight greater than or equal to (>=) 50 kilogram (kg) and body mass index (BMI) within the range 19-29.9 kilogram per meter square (kg/m2) (inclusive).
* Male participants are eligible to participate in the study.
* A female participant is eligible to participate if she is not pregnant or breastfeeding or using highly effective contraceptive methods. Woman of non-childbearing potential can also participate.
* A sensitive pregnancy test is required to be negative on the day of each challenge.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Significant history of or current, cardiovascular (including hypotension, severe hypertension, vasomotor instability), respiratory (including asthma), renal, gastrointestinal, endocrine, hematological, infectious or neurological disorders constituting a risk when taking part in the study or interfering with the interpretation of data.
* History or presence of significant skin disorder (such as but not limited to chronic urticaria, atopic dermatitis, severe eczema, psoriasis or skin cancer).
* History of risk for or actual experience of complications from skin biopsy including excess bleeding, infection, or scarring/keloid formation.
* Abnormal blood pressure as determined by the investigator.
* Alanine transaminase (ALT) >1.5 times upper limit of normal (ULN).
* Total bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if total bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 millisecond (msec), based on the mean of triplicate ECGs.
* Use of any form of H1 or H2 antihistamine, tricyclic antidepressants, beta2 agonists, dopamine, or beta blocking agents within 14 days before the first challenge visit through final assessments.
* Use of topical medications such as but not limited to retinoids, steroids, and transdermal hormone replacement therapies on or near the intended site of application within 8 weeks prior to dosing through treatment follow up. Use of other topical preparations such as those containing vitamins, supplements or herbal within 2 weeks prior to dosing through treatment follow up.
* Past or intended use of any other non-topical over-the-counter or prescription medication, including herbal medications, within 7 days before the first challenge visit, unless, in the opinion of the investigator and GlaxoSmithKline medical monitor, the medication will not constitute a risk when taking the study intervention or interfere with the interpretation of data.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 3 months.
* Current enrolment in any clinical study involving an investigational study intervention or any other type of medical research.
* Current enrolment or past participation in this study.
* Presence of Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HbcAb) at screening or within 3 months before the first challenge day.
* Positive Hepatitis C antibody test result at screening or within 3 months before the first challenge day.
* Positive Hepatitis C RNA test result at screening or within 3 months before the first challenge day.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test at screening or within 3 months before the first challenge day.
* Current use of known drugs of abuse.
* Participants who present with damaged skin including sunburn, scar tissue, moles, uneven skin tones and dark skin tone (Fitzpatrick>2), tattoos, body piercings, branding or other skin disfiguration on or near the intended site of application which could interfere with the assessments
* Regular alcohol consumption within 6 months before the study defined as an average weekly intake of >21 units for males or >14 units for females.
* Smoking test result indicative of smoking, history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Unable to refrain from the use of topical medications from before the first to after the last challenge visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Background] Ten Voorde W, Akinseye C, Abdisalaam I, Wind S, Klarenbeek N, Bergmans M, van Doorn M, Rissmann R, Kaur R, Hotee S, Foster K, Nair A, Fortunato L, Macphee C, Mole S, Baumann K, Brigandi R. Intradermal substance P as a challenge agent in healthy individuals. Clin Transl Sci. 2023 Oct;16(10):1856-1865. doi: 10.1111/cts.13592. Epub 2023 Aug 7. PMID 37547990

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, 2-part, sequential, prospective enabling study of Substance P (SP) intradermal challenge in healthy participants conducted at a single center in the Netherlands.
Pre-assignment Details: A total of 32 participants were enrolled (Enrolled population: All participants in the screened population who entered the study) in Part 1 (12 participants) and Part 2 (20 participants) of the study.
Groups:
- Part 1- Skin Challenges: Healthy participants were first administered saline, by intradermal injection, and histamine by skin prick, as negative and positive controls. Participants with acceptable saline and histamine responses, were administered up to 4 intradermal injections of Substance P sequentially from lowest to highest concentration (5, 15, 50, 150 and 500 picomole [PMOL]) at challenge visit 1 (Day 1) and wheal and flare responses were assessed. There was no Challenge Visit 2 in Part 1.
- Part 1- No Skin Challenges: Healthy participants were first administered saline, by intradermal injection, and histamine by skin prick, as negative and positive controls. Participants whose wheal responses did not meet the acceptable saline and histamine response within 20 minutes of each control challenge or who were withdrawn from the study, independent of the wheal response acceptability, were not administered Substance P.
- Part 2- Skin Challenges: Healthy participants were first administered saline, by intradermal injection, and histamine by skin prick, as negative and positive controls. Participants with acceptable saline and histamine responses were administered up to 4 intradermal injections of Substance P sequentially from lowest to highest concentration (5, 15, 50 and 150 PMOL) and wheal and flare responses were assessed along with Intradermal microdialysis (IDM) after Challenge Visit 1 (Day 1). At Challenge Visit 2 (Week 2), participants were administered up to 6 Substance P intradermal injections and wheal and flare response, IDM and biopsies were taken (one from each challenged site and one from a non-challenged area of skin.
Period: Part 1 (Up to Day 1)
Arm/Group | Part 1- Skin Challenges | Part 1- No Skin Challenges | Part 2- Skin Challenges
Started | 9 | 3 | 0
Number of Participants Who Received SP 5 PMOL | 9 | 0 | 0
Number of Participants Who Received SP 15 PMOL | 9 | 0 | 0
Number of Participants Who Received SP 50 PMOL | 4 | 0 | 0
Number of Participants Who Received SP 150 PMOL | 9 | 0 | 0
Number of Participants Who Received SP 500 PMOL | 5 | 0 | 0
Completed | 9 | 0 | 0
Not Completed | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Part 2 (Up to 3 Weeks)
Arm/Group | Part 1- Skin Challenges | Part 1- No Skin Challenges | Part 2- Skin Challenges
Started | 0 | 0 | 20
Number of Participants Who Received SP 5 PMOL | 0 | 0 | 20
Number of Participants Who Received SP 15 PMOL | 0 | 0 | 20
Number of Participants Who Received SP 50 PMOL | 0 | 0 | 20
Number of Participants Who Received SP 150 PMOL | 0 | 0 | 20
Completed | 0 | 0 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for Enrolled population which consisted of all participants in the screened population who entered the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1- Skin Challenges | Part 1- No Skin Challenges | Part 2- Skin Challenges | Total
Number analyzed (Participants) | 9 | 3 | 20 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.0 (3.50) | 22.0 (4.58) | 26.8 (9.34) | 25.3 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 13 | 20
  Male | 3 | 2 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White- Arabic / North African Heritage | 0 | 0 | 2 | 2
  White- White/ Caucasian/ European Heritage | 9 | 3 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Wheal Response-time Area Under the Curve (AUC) Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1)
Description: Wheal response-time AUC during the 2 hours post-challenge period following skin challenge for Substance P (SP) was calculated using the trapezoidal rule. The wheal response was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50, 150 and 500 picomoles (pmol) during the 2 hours post-challenge period.
Time Frame: 0, 5, 10, 15, 20, 40, 60, 90 and 120 minutes post-challenge on Day 1 (Visit 1)
Population: Safety Population consisted of all participants in the enrolled analysis set who received at least one challenge-related study procedure on their (first) challenge day. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter square*minutes
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Millimeter square*minutes
  Saline | 155.2379 (97.43852)
  Histamine | 2151.2320 (1352.66124)
  SP 5 pmol | 2749.0997 (2000.66201)
  SP 15 pmol | 5727.2220 (3859.78704)
  SP 50 pmol: number analyzed (Participants) | 4
  SP 50 pmol | 7111.5570 (5388.48885)
  SP 150 pmol | 8295.6310 (5912.58152)
  SP 500 pmol: number analyzed (Participants) | 5
  SP 500 pmol | 12540.9840 (14705.68961)

2. Primary Outcome: Part 2: Wheal Response-time AUC Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: Wheal response-time AUC during the 2 hours post-challenge period following skin challenge for Substance P was calculated using the trapezoidal rule. The wheal response was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50 and 150 pmol during the 2 hours post-challenge period.
Time Frame: 0, 5, 10, 15, 20, 30, 40, 60, 90 and 120 minutes post-challenge on Day 1 (Visit 1) and on Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter square*minutes
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Millimeter square*minutes
  Saline: 2 hours post-challenge on Day 1 | 157.9157 (110.11185)
  Saline: 2 hours post-challenge at Week 2 | 216.5196 (113.81519)
  Histamine: 2 hours post-challenge on Day 1 | 2617.3622 (1362.88319)
  Histamine: 2 hours post-challenge at Week 2 | 2486.9477 (1171.55762)
  SP 5 pmol: 2 hours post-challenge on Day 1 | 4534.4513 (2153.69897)
  SP 5 pmol: 2 hours post-challenge at Week 2 | 4563.5113 (2517.52789)
  SP 15 pmol: 2 hours post-challenge on Day 1 | 6754.7067 (3501.44122)
  SP 15 pmol: 2 hours post-challenge at Week 2 | 6506.0915 (3199.02966)
  SP 50 pmol: 2 hours post-challenge on Day 1 | 8937.9117 (4089.24955)
  SP 50 pmol: 2 hours post-challenge at Week 2 | 9763.2271 (4963.46223)
  SP 150 pmol:2 hours post-challenge on Day 1 | 11017.5544 (4779.69981)
  SP 150 pmol: 2 hours post-challenge at Week 2 | 9977.7777 (4155.85567)

3. Secondary Outcome: Part 1: Maximum Observed Wheal Area Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1)
Description: Wheal area was calculated using the following formula: 1/4 * pi * longest diameter * orthogonal diameter, for area of an ellipse, using the longest and orthogonal diameters measured by the calliper method. The maximum observed wheal area was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50, 150 and 500 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter square
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Millimeter square
  Saline | 15.2152 (8.97791)
  Histamine | 44.5782 (16.73404)
  SP 5 pmol | 42.4284 (20.26132)
  SP 15 pmol | 82.7571 (41.76154)
  SP 50 pmol: number analyzed (Participants) | 4
  SP 50 pmol | 99.8398 (48.06381)
  SP 150 pmol | 126.1186 (55.28040)
  SP 500 pmol: number analyzed (Participants) | 5
  SP 500 pmol | 194.0748 (178.88175)

4. Secondary Outcome: Part 2: Maximum Observed Wheal Area Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P Across- at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: Wheal area was calculated using the following formula: 1/4 * pi * longest diameter * orthogonal diameter, for area of an ellipse, using the longest and orthogonal diameters measured by the calliper method. The maximum observed wheal area was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50 and 150 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1) and 2 hours post-challenge at Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter square
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Millimeter square
  Saline : 2 hours post-challenge on Day 1 | 16.6335 (11.36559)
  Saline: 2 hours post-challenge at Week 2 | 21.7610 (12.79723)
  Histamine: 2 hours post-challenge on Day 1 | 53.1929 (26.57857)
  Histamine: 2 hours post-challenge at Week 2 | 52.8665 (16.31003)
  SP 5 pmol: 2 hours post-challenge on Day 1 | 85.8111 (23.45193)
  SP 5 pmol: 2 hours post-challenge at Week 2 | 92.1595 (24.44909)
  SP 15 pmol: 2 hours post-challenge on Day 1 | 112.9690 (30.79242)
  SP 15 pmol: 2 hours post-challenge at Week 2 | 113.0940 (26.92327)
  SP 50 pmol: 2 hours post-challenge on Day 1 | 134.6049 (39.38378)
  SP 50 pmol: 2 hours post-challenge at Week 2 | 151.1447 (39.31424)
  SP 150 pmol:2 hours post-challenge on Day 1 | 148.8571 (47.72791)
  SP 150 pmol: 2 hours post-challenge at Week 2 | 153.0084 (39.81310)

5. Secondary Outcome: Part 1: Time to Maximum Observed Wheal Area Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1)
Description: Time to maximum observed wheal area was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50, 150 and 500 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Minutes
  Saline | 5.0 [5 to 11]
  Histamine | 20.0 [15 to 42]
  SP 5 pmol | 20.0 [5 to 60]
  SP 15 pmol | 20.0 [10 to 40]
  SP 50 pmol: number analyzed (Participants) | 4
  SP 50 pmol | 17.5 [10 to 21]
  SP 150 pmol | 20.0 [10 to 60]
  SP 500 pmol: number analyzed (Participants) | 5
  SP 500 pmol | 20.0 [5 to 20]

6. Secondary Outcome: Part 2: Time to Maximum Observed Wheal Area Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: Time to maximum observed wheal area was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50 and 150 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1) and 2 hours post-challenge at Week 2 (Visit 2)
Population: Safety Population
Measure: Median (Full Range); unit: Minutes
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Minutes
  Saline : 2 hours post-challenge on Day 1 | 5.0 [4 to 10]
  Saline: 2 hours post-challenge at Week 2 | 5.0 [4 to 10]
  Histamine: 2 hours post-challenge on Day 1 | 30.0 [9 to 62]
  Histamine: 2 hours post-challenge at Week 2 | 24.5 [14 to 60]
  SP 5 pmol: 2 hours post-challenge on Day 1 | 18.5 [9 to 39]
  SP 5 pmol: 2 hours post-challenge at Week 2 | 19.0 [9 to 39]
  SP 15 pmol: 2 hours post-challenge on Day 1 | 19.5 [8 to 90]
  SP 15 pmol: 2 hours post-challenge at Week 2 | 18.5 [11 to 89]
  SP 50 pmol: 2 hours post-challenge on Day 1 | 23.5 [4 to 60]
  SP 50 pmol: 2 hours post-challenge at Week 2 | 25.0 [15 to 59]
  SP 150 pmol:2 hours post-challenge on Day 1 | 28.0 [5 to 90]
  SP 150 pmol: 2 hours post-challenge at Week 2 | 27.5 [15 to 41]

7. Secondary Outcome: Part 1: Time to Complete Wheal Area Disappearance Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1)
Description: Time to complete wheal area disappearance was calculated during the 2 hours post-challenge period. Complete disappearance is defined as a value of 0 for wheal area, longest diameter or orthogonal diameter. Participants who did not have a disappearance within the 2 hours post challenge period were excluded. Time to complete wheal area disappearance was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50, 150 and 500 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Minutes
  Saline | 39.0 [15 to 55]
  Histamine | 90.0 [56 to 93]
  SP 5 pmol: number analyzed (Participants) | 7
  SP 5 pmol | 62.0 [40 to 120]
  SP 15 pmol: number analyzed (Participants) | 7
  SP 15 pmol | 120.0 [42 to 121]
  SP 50 pmol: number analyzed (Participants) | 2
  SP 50 pmol | 74.5 [59 to 90]
  SP 150 pmol: number analyzed (Participants) | 6
  SP 150 pmol | 75.5 [40 to 120]
  SP 500 pmol: number analyzed (Participants) | 4
  SP 500 pmol | 104.5 [60 to 120]

8. Secondary Outcome: Part 2: Time to Complete Wheal Area Disappearance Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: Time to complete wheal area disappearance was calculated during the 2 hours post-challenge period. Complete disappearance is defined as a value of 0 for wheal area, longest diameter or orthogonal diameter. Participants who did not have a disappearance within the 2 hours post challenge period were excluded. Time to complete wheal area disappearance was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50 and 150 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1) and 2 hours post-challenge at Week 2 (Visit 2)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Minutes
  Saline : 2 hours post-challenge on Day 1 | 16.0 [11 to 30]
  Saline: 2 hours post-challenge at Week 2 | 20.0 [11 to 27]
  Histamine: 2 hours post-challenge on Day 1 | 90.5 [6 to 120]
  Histamine: 2 hours post-challenge at Week 2: number analyzed (Participants) | 19
  Histamine: 2 hours post-challenge at Week 2 | 90.0 [40 to 120]
  SP 5 pmol: 2 hours post-challenge on Day 1 | 89.0 [38 to 121]
  SP 5 pmol: 2 hours post-challenge at Week 2: number analyzed (Participants) | 19
  SP 5 pmol: 2 hours post-challenge at Week 2 | 61.0 [58 to 121]
  SP 15 pmol: 2 hours post-challenge on Day 1: number analyzed (Participants) | 18
  SP 15 pmol: 2 hours post-challenge on Day 1 | 90.0 [38 to 121]
  SP 15 pmol: 2 hours post-challenge at Week 2: number analyzed (Participants) | 19
  SP 15 pmol: 2 hours post-challenge at Week 2 | 88.0 [40 to 123]
  SP 50 pmol: 2 hours post-challenge on Day 1: number analyzed (Participants) | 16
  SP 50 pmol: 2 hours post-challenge on Day 1 | 90.0 [58 to 121]
  SP 50 pmol: 2 hours post-challenge at Week 2: number analyzed (Participants) | 19
  SP 50 pmol: 2 hours post-challenge at Week 2 | 90.0 [60 to 122]
  SP 150 pmol:2 hours post-challenge on Day 1: number analyzed (Participants) | 16
  SP 150 pmol:2 hours post-challenge on Day 1 | 104.5 [59 to 121]
  SP 150 pmol: 2 hours post-challenge at Week 2: number analyzed (Participants) | 19
  SP 150 pmol: 2 hours post-challenge at Week 2 | 90.0 [60 to 121]

9. Secondary Outcome: Part 1: Flare Response-time AUC Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1)
Description: Flare response-time AUC during the 2 hours post-challenge period following skin challenge for Substance P was calculated using the trapezoidal rule. The flare response was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50, 150 and 500 pmol during the 2 hours post-challenge period.
Time Frame: 0, 5, 10, 15, 20, 40, 60, 90 and 120 minutes post-challenge on Day 1 (Visit 1)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed. Zeros reported reflect measured data derived during analysis.
Measure: Mean (Standard Deviation); unit: Millimeter square*minutes
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Millimeter square*minutes
  Saline | 0.0000 (0.00000)
  Histamine | 47977.8047 (35779.56892)
  SP 5 pmol | 8232.5351 (10307.53738)
  SP 15 pmol | 26562.8609 (22150.49500)
  SP 50 pmol: number analyzed (Participants) | 4
  SP 50 pmol | 53505.6580 (31081.10933)
  SP 150 pmol | 54407.2697 (34805.98795)
  SP 500 pmol: number analyzed (Participants) | 5
  SP 500 pmol | 64978.5132 (67350.94024)

10. Secondary Outcome: Part 2: Flare Response-time AUC Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: Flare response-time AUC during the 2 hours post-challenge period following skin challenge for Substance P was calculated using the trapezoidal rule. The flare response variable was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50 and 150 pmol during the 2 hours post-challenge period.
Time Frame: 0, 5, 10, 15, 20, 30, 40, 60, 90 and 120 minutes post-challenge on Day 1 (Visit 1) and on Week 2 (Visit 2)
Population: Safety Population. Zeros reported reflect measured data derived during analysis.
Measure: Mean (Standard Deviation); unit: Millimeter square*minutes
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Millimeter square*minutes
  Saline : 2 hours post-challenge on Day 1 | 0.0000 (0.00000)
  Saline: 2 hours post-challenge at Week 2 | 0.0000 (0.00000)
  Histamine: 2 hours post-challenge on Day 1 | 42825.0421 (31599.99246)
  Histamine: 2 hours post-challenge at Week 2 | 50717.6974 (35294.02927)
  SP 5 pmol: 2 hours post-challenge on Day 1 | 20515.8733 (17779.84450)
  SP 5 pmol: 2 hours post-challenge at Week 2 | 30689.5773 (29415.10538)
  SP 15 pmol: 2 hours post-challenge on Day 1 | 48796.3715 (31253.62644)
  SP 15 pmol: 2 hours post-challenge at Week 2 | 52359.5705 (34531.05693)
  SP 50 pmol: 2 hours post-challenge on Day 1 | 68798.6958 (36263.19533)
  SP 50 pmol: 2 hours post-challenge at Week 2 | 81245.6716 (50591.14135)
  SP 150 pmol:2 hours post-challenge on Day 1 | 76360.0164 (32955.71419)
  SP 150 pmol: 2 hours post-challenge at Week 2 | 77243.2496 (37747.18154)

11. Secondary Outcome: Part 1: Maximum Observed Flare Area Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1)
Description: Flare area was calculated using the following formula: 1/4 * pi * longest diameter * orthogonal diameter, for area of an ellipse, using the longest and orthogonal diameters measured by the calliper method. The maximum observed flare area was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50, 150 and 500 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimeter square
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Millimeter square
  Saline | 0.0000 (0.00000)
  Histamine | 1209.6224 (604.47133)
  SP 5 pmol | 619.6359 (940.26080)
  SP 15 pmol | 1422.8103 (763.79695)
  SP 50 pmol: number analyzed (Participants) | 4
  SP 50 pmol | 2240.1860 (971.83781)
  SP 150 pmol | 2282.5890 (1149.03190)
  SP 500 pmol: number analyzed (Participants) | 5
  SP 500 pmol | 2383.3822 (1590.27531)

12. Secondary Outcome: Part 2: Maximum Observed Flare Area Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P Across- at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: Flare area was calculated using the following formula: 1/4 * pi * longest diameter * orthogonal diameter, for area of an ellipse, using the longest and orthogonal diameters measured by the calliper method. The maximum observed flare area was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50 and 150 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1) and 2 hours post-challenge At Week 2 (Visit 2)
Population: Safety Population. Zeros reported reflect measured data derived during analysis.
Measure: Mean (Standard Deviation); unit: Millimeter square
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Millimeter square
  Saline : 2 hours post-challenge on Day 1 | 0.0000 (0.00000)
  Saline: 2 hours post-challenge at Week 2 | 0.0000 (0.00000)
  Histamine: 2 hours post-challenge on Day 1 | 1110.0748 (514.76131)
  Histamine: 2 hours post-challenge at Week 2 | 1392.6911 (671.10955)
  SP 5 pmol: 2 hours post-challenge on Day 1 | 1035.4156 (572.41049)
  SP 5 pmol: 2 hours post-challenge at Week 2 | 1398.2891 (1007.58015)
  SP 15 pmol: 2 hours post-challenge on Day 1 | 1892.5393 (791.10820)
  SP 15 pmol: 2 hours post-challenge at Week 2 | 1956.0858 (1018.31529)
  SP 50 pmol: 2 hours post-challenge on Day 1 | 2229.9920 (772.48097)
  SP 50 pmol: 2 hours post-challenge at Week 2 | 2575.5958 (1627.22854)
  SP 150 pmol:2 hours post-challenge on Day 1 | 2058.1909 (660.32625)
  SP 150 pmol: 2 hours post-challenge at Week 2 | 2281.9739 (853.10184)

13. Secondary Outcome: Part 1: Time to Maximum Observed Flare Area Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1)
Description: Time to maximum observed flare area was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50, 150 and 500 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Minutes
  Saline | 5.0 [4 to 5]
  Histamine | 15.0 [5 to 21]
  SP 5 pmol | 10.0 [5 to 11]
  SP 15 pmol | 5.0 [5 to 10]
  SP 50 pmol: number analyzed (Participants) | 4
  SP 50 pmol | 5.0 [4 to 5]
  SP 150 pmol | 6.0 [5 to 15]
  SP 500 pmol: number analyzed (Participants) | 5
  SP 500 pmol | 5.0 [5 to 5]

14. Secondary Outcome: Part 2: Time to Maximum Observed Flare Area Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: Time to maximum observed flare area was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50 and 150 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1) and 2 hours post-challenge At Week 2 (Visit 2)
Population: Safety Population
Measure: Median (Full Range); unit: Minutes
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Minutes
  Saline : 2 hours post-challenge on Day 1 | 5.0 [4 to 6]
  Saline: 2 hours post-challenge at Week 2 | 5.0 [4 to 6]
  Histamine: 2 hours post-challenge on Day 1 | 11.0 [5 to 30]
  Histamine: 2 hours post-challenge at Week 2 | 6.0 [5 to 20]
  SP 5 pmol: 2 hours post-challenge on Day 1 | 5.0 [4 to 14]
  SP 5 pmol: 2 hours post-challenge at Week 2 | 5.0 [5 to 18]
  SP 15 pmol: 2 hours post-challenge on Day 1 | 5.0 [4 to 15]
  SP 15 pmol: 2 hours post-challenge at Week 2 | 5.0 [4 to 15]
  SP 50 pmol: 2 hours post-challenge on Day 1 | 5.0 [3 to 15]
  SP 50 pmol: 2 hours post-challenge at Week 2 | 5.5 [4 to 20]
  SP 150 pmol:2 hours post-challenge on Day 1 | 5.0 [4 to 16]
  SP 150 pmol: 2 hours post-challenge at Week 2 | 5.0 [4 to 19]

15. Secondary Outcome: Part 1: Time to Complete Flare Area Disappearance Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1)
Description: Time to complete flare area disappearance was calculated during the 2 hours post-challenge period. Complete disappearance is defined as a value of 0 for flare area, longest diameter or orthogonal diameter. Participants who did not have a disappearance within the 2 hours post challenge period were excluded. Time to complete wheal area disappearance was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50, 150 and 500 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Minutes
  Saline | 5.0 [4 to 5]
  Histamine | 89.0 [56 to 93]
  SP 5 pmol | 20.0 [10 to 60]
  SP 15 pmol | 42.0 [19 to 90]
  SP 50 pmol: number analyzed (Participants) | 4
  SP 50 pmol | 59.5 [41 to 90]
  SP 150 pmol | 60.0 [40 to 90]
  SP 500 pmol: number analyzed (Participants) | 5
  SP 500 pmol | 61.0 [20 to 90]

16. Secondary Outcome: Part 2: Time to Complete Flare Area Disappearance Over the 2 Hours Post-challenge Period Following Skin Challenge With Substance P- at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: Time to complete flare area disappearance was calculated during the 2 hours post-challenge period. Complete disappearance is defined as a value of 0 for wheal area, longest diameter or orthogonal diameter. Participants who did not have a disappearance within the 2 hours post challenge period were excluded. Time to complete wheal area disappearance was calculated for each control challenge (saline and histamine) and each ascending Substance P concentration: 5, 15, 50 and 150 pmol during the 2 hours post-challenge period.
Time Frame: 2 hours post-challenge on Day 1 (Visit 1) and 2 hours post-challenge At Week 2 (Visit 2)
Population: Safety Population
Measure: Median (Full Range); unit: Minutes
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Minutes
  Saline : 2 hours post-challenge on Day 1 | 5.0 [4 to 6]
  Saline: 2 hours post-challenge at Week 2 | 5.0 [4 to 6]
  Histamine: 2 hours post-challenge on Day 1 | 75.5 [39 to 119]
  Histamine: 2 hours post-challenge at Week 2 | 76.0 [39 to 94]
  SP 5 pmol: 2 hours post-challenge on Day 1 | 40.0 [5 to 60]
  SP 5 pmol: 2 hours post-challenge at Week 2 | 39.0 [6 to 89]
  SP 15 pmol: 2 hours post-challenge on Day 1 | 59.0 [13 to 89]
  SP 15 pmol: 2 hours post-challenge at Week 2 | 59.0 [15 to 88]
  SP 50 pmol: 2 hours post-challenge on Day 1 | 61.0 [29 to 91]
  SP 50 pmol: 2 hours post-challenge at Week 2 | 60.0 [30 to 91]
  SP 150 pmol:2 hours post-challenge on Day 1 | 90.0 [29 to 91]
  SP 150 pmol: 2 hours post-challenge at Week 2 | 88.0 [40 to 91]

17. Secondary Outcome: Part 1: Number of Participants With Non-serious Adverse Events (AEs) and Serious AEs (SAEs)- Substance P Only
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with non-serious AEs and SAEs is presented.
Time Frame: Up to Day 1
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Participants
  Non-serious AEs | 1
  SAEs | 0

18. Secondary Outcome: Part 2: Number of Participants With Non-serious AEs and SAEs- Substance P Only
Description: as for outcome 17
Time Frame: Up to 3 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Participants
  Non-serious AEs | 2
  SAEs | 0

19. Secondary Outcome: Part 1: Number of Participants With Worst Case Vital Signs Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline- Substance P Only at Challenge Visit 1 (Day 1)
Description: Vital signs parameters including Systolic blood pressure (SBP), Diastolic blood pressure (DBP) and heart rate were measured in a semi-supine position after 5 minutes of rest with a completely automated device. PCI ranges were: SBP (Lower: less than [<]85 and Upper: greater than [>]160 millimeters of mercury [mmHg]); DBP (Lower: <45 and Upper: >100 mmHg); Heart Rate: (Lower: <40 and Upper: >110 beats per minute). Baseline value is defined as the latest non-missing pre-first control challenge assessment value at challenge visit 1, including those from unscheduled visits. Participants were counted in the worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages (%) may not add to 100%.
Time Frame: At Day 1 (Visit 1)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Participants
  SBP: To low | 0
  SBP: To within range or no Change | 9
  SBP: To High | 0
  DBP: To low | 0
  DBP: To within range or no Change | 9
  DBP: To High | 0
  Heart rate: To low | 0
  Heart rate: To within range or no Change | 9
  Heart rate: To High | 0

20. Secondary Outcome: Part 2: Number of Participants With Worst Case Vital Signs Parameter Results by Potential Clinical Importance (PCI) Post-Baseline Relative to Baseline- Substance P Only at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: Vital signs parameters including SBP, DBP and heart rate were measured in a semi-supine position after 5 minutes of rest with a completely automated device. PCI ranges were: SBP (Lower: <85 and Upper: >160 mmHg); DBP (Lower: <45 and Upper: >100 mmHg); Heart Rate: (Lower: <40 and Upper: >110 beats per minute). Baseline value is defined as the latest non-missing pre-first control challenge assessment value at challenge visit 1 and challenge visit 2, including those from unscheduled visits. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Participants were counted in the worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants were counted twice if the participant had values that changed "To Low" and "To High", so the % may not add to 100%.
Time Frame: At Day 1 (Visit 1) and Week 2 (Visit 2)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Participants
  SBP: To low, Day 1 | 0
  SBP: To within range or no Change, Day 1 | 20
  SBP: To High, Day 1 | 0
  SBP: To low, Week 2 | 0
  SBP: To within range or no Change, Week 2 | 20
  SBP: To High, Week 2 | 0
  DBP: To low, Day 1 | 0
  DBP: To within range or no Change, Day 1 | 20
  DBP: To High, Day 1 | 0
  DBP: To low, Week 2 | 0
  DBP: To within range or no Change, Week 2 | 20
  DBP: To High, Week 2 | 0
  Heart rate: To low, Day 1 | 0
  Heart rate: To within range or no Change, Day 1 | 20
  Heart rate: To High, Day 1 | 0
  Heart rate: To low, Week 2 | 0
  Heart rate: To within range or no Change,Week 2 | 20
  Heart rate: To High, Week 2 | 0

21. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophil Count, Platelet Count and White Blood Cell Count- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of hematology parameters: basophils, eosinophils, lymphocytes, monocytes, total neutrophil count, platelet count and white blood cell count. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Giga cells per liter
  Basophils | 0.041 (0.0215)
  Eosinophils | 0.112 (0.1402)
  Lymphocytes | 1.818 (0.3138)
  Monocytes | 0.413 (0.1055)
  Total neutrophil count | 3.141 (1.1766)
  Platelet count | 256.8 (56.77)
  White blood cell count | 5.526 (1.3657)

22. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophil Count, Platelet Count and White Blood Cell Count- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of hematology parameters: Basophils, eosinophils, lymphocytes, monocytes, total neutrophil count, platelet count and white blood cell count. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Giga cells per liter
  Basophils | 0.045 (0.0235)
  Eosinophils | 0.308 (0.3889)
  Lymphocytes | 2.016 (0.5291)
  Monocytes | 0.490 (0.1649)
  Total neutrophil count | 3.788 (1.3756)
  Platelet count | 244.5 (54.47)
  White blood cell count | 6.646 (1.7007)

23. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hemoglobin- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of hematology parameter: Hemoglobin. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Grams per liter | 140.186580 (11.4507222)

24. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hemoglobin- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of hematology parameter: Hemoglobin. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Grams per liter | 133.821787 (8.9711806)

25. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hematocrit- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of hematology parameter: Hematocrit. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Proportion of red blood cells in blood | 0.4117 (0.02807)

26. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hematocrit- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of hematology parameter: Hematocrit. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Proportion of red blood cells in blood | 0.3929 (0.02349)

27. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Mean Corpuscle Hemoglobin- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of hematology parameter: Mean corpuscle hemoglobin. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Picograms | 30.203673 (1.0991155)

28. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Mean Corpuscle Hemoglobin- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of hematology parameter: Mean corpuscle hemoglobin. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Picograms | 30.204568 (1.6675822)

29. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Mean Corpuscle Volume- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of hematology parameter: Mean corpuscle volume. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Femtoliters | 89.0 (4.09)

30. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Mean Corpuscle Volume- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of hematology parameter: Mean corpuscle volume. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Femtoliters | 88.7 (2.92)

31. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Red Blood Cell Count- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of hematology parameter: Red blood cell count. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Trillion cells per liter | 4.652 (0.5003)

32. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Red Blood Cell Count- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of hematology parameter: Red blood cell count. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Trillion cells per liter | 4.440 (0.3345)

33. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Reticulocyte- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of hematology parameter: Reticulocyte. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 7
Percentage of reticulocytes | 0.01197 (0.002160)

34. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Reticulocyte- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of hematology parameter: Reticulocyte. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Percentage of reticulocytes | 0.01482 (0.004017)

35. Secondary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Alkaline Phosphatase, Alanine Aminotransferase and Aspartate Aminotransferase- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of clinical chemistry parameters: Alkaline phosphatase, alanine aminotransferase and aspartate aminotransferase. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
International units per liter
  Alkaline phosphatase | 71.1 (18.38)
  Alanine aminotransferase | 19.0 (8.82)
  Aspartate aminotransferase | 18.8 (3.70)

36. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: Alkaline Phosphatase, Alanine Aminotransferase and Aspartate Aminotransferase- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of clinical chemistry parameters: Alkaline phosphatase, alanine aminotransferase and aspartate aminotransferase. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
International units per liter
  Alkaline phosphatase | 72.4 (30.54)
  Alanine aminotransferase | 19.7 (7.38)
  Aspartate aminotransferase | 21.1 (5.85)

37. Secondary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Total Bilirubin and Creatinine- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of clinical chemistry parameters: Total Bilirubin and creatinine. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Micromoles per liter
  Total bilirubin | 11.6 (3.50)
  Creatinine | 60.3 (10.54)

38. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: Total Bilirubin and Creatinine- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of clinical chemistry parameters: Total bilirubin and creatinine. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Micromoles per liter
  Total bilirubin | 6.7 (2.80)
  Creatinine | 66.9 (13.67)

39. Secondary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Calcium, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN)- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of clinical chemistry parameters: Calcium, glucose, potassium, sodium, and urea/BUN. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Millimoles per liter
  Calcium | 2.350 (0.0910)
  Glucose | 5.09 (0.457)
  Potassium | 4.27 (0.265)
  Sodium | 141.8 (1.86)
  Urea/BUN | 4.04 (0.979)

40. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: Calcium, Glucose, Potassium, Sodium, and Urea/BUN- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of clinical chemistry parameters: Calcium, glucose, potassium, sodium, and urea/BUN. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Millimoles per liter
  Calcium | 2.346 (0.1074)
  Glucose | 4.89 (0.713)
  Potassium | 4.19 (0.315)
  Sodium | 141.1 (2.38)
  Urea/BUN | 4.38 (1.614)

41. Secondary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameter: Total Protein- Substance P Only at Challenge Visit 1 (Day 1)
Description: Blood samples were collected for the analysis of clinical chemistry parameter: Total protein. Baseline value is defined as the latest non-missing pre-first control challenge assessment value (Within 1 hour before first control challenge) at challenge visit 1, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Day 1 (Visit 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Grams per liter | 69.4 (3.97)

42. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameter: Total Protein- Substance P Only at Challenge Visit 2 (Week 2)
Description: Blood samples were collected for the analysis of clinical chemistry parameter: Total protein. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1: pre-dose) and At Week 2 (Visit 2)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Grams per liter | 68.8 (3.72)

43. Secondary Outcome: Part 1: Number of Participants With Worst Case Urinalysis Parameters Post-Baseline Relative to Baseline- Substance P Only at Challenge Visit 1 (Day 1)
Description: Urine samples were collected for the analysis of urinalysis parameters: Occult blood, glucose, ketones and protein by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters indicate proportional concentrations in the urine sample. Number of participants with abnormal results were reported as 'Any increase' if there was any increase in their urine concentrations compared to Baseline. Participants whose value was unchanged or whose value was decreased, were recorded in the 'No change/Decreased' category. Baseline value is defined as the latest non-missing pre-first control challenge assessment value at challenge visit 1, including those from unscheduled visits.
Time Frame: At Day 1 (Visit 1)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Participants
  Occult blood: No change/decreased | 8
  Occult blood: Any increase | 1
  Glucose: No change/decreased | 9
  Glucose: Any increase | 0
  Ketones No change/decreased | 9
  Ketones: Any increase | 0
  Protein: No change/decreased | 9
  Protein: Any increase | 0

44. Secondary Outcome: Part 2: Number of Participants With Worst Case Urinalysis Parameters Post-Baseline Relative to Baseline- Substance P Only at Challenge Visit 2 (Week 2)
Description: Urine samples were collected for the analysis of urinalysis parameters: Occult blood, glucose, ketones and protein by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters indicate proportional concentrations in the urine sample. Number of participants with abnormal results were reported as 'Any increase' if there was any increase in their urine concentrations compared to Baseline. Participants whose value was unchanged or whose value was decreased, were recorded in the 'No change/Decreased' category. For Part 2, the Baseline for Visit 2 is defined as the latest assessment performed after Visit 1 visits (such as Unscheduled) but before the first Visit 2 challenge.
Time Frame: At Week 2 (Visit 2)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Participants
  Occult blood: No change/decreased | 20
  Occult blood: Any increase | 0
  Glucose: No change/decreased | 20
  Glucose: Any increase | 0
  Ketones No change/decreased | 20
  Ketones: Any increase | 0
  Protein: No change/decreased | 20
  Protein: Any increase | 0

45. Secondary Outcome: Part 1: Number of Participants With Clinically Significant Abnormal 12-lead Electrocardiogram (ECG) Findings- Substance P Only at Challenge Visit 1 (Day 1)
Description: 12-lead ECGs were obtained by using an automated ECG machine that measured PR, QRS, QT, and corrected QT (QTc) intervals and calculated heart rate. Data for abnormal, clinically significant (CS) ECG findings are presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: At Day 1 (Visit 1)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1- Skin Challenges
Number analyzed (Participants) | 9
Participants | 0

46. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Abnormal 12-lead ECG Findings- Substance P Only at Challenge Visit 1 (Day 1) and Challenge Visit 2 (Week 2)
Description: 12-lead ECGs were obtained by using an automated ECG machine that measured PR, QRS, QT, and QTc intervals and calculated heart rate. Data for abnormal, CS ECG findings are presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: At Day 1 (Visit 1) and Week 2 (Visit 2)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2- Skin Challenges
Number analyzed (Participants) | 20
Participants
  Day 1 | 0
  Week 2 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-serious AEs were collected from the start of study treatment up to Day 1 for Part 1 and Up to Week 3 for Part 2.
Description: SAEs and Non-SAEs were reported for the Safety Population which comprised of all participants in the enrolled analysis set who received at least one challenge-related study procedure on their (first) challenge day. AEs were not collected for "Part 1:No Skin Challenges" arm (N=3), as they did not receive any challenge related study procedure, hence were not included in Safety population.
Arm/Group | Part 1- Skin Challenges | Part 2- Skin Challenges
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/20
Other Adverse Events (participants affected / at risk) | 1/9 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1- Skin Challenges (N=9) | Part 2- Skin Challenges (N=20)
Headache (Nervous system disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT04676763/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT04676763/SAP_001.pdf